CLINICAL TRIAL: NCT05054764
Title: Promus PREMIER Below The Knee Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sengkang General Hospital (Other)
Responsible Party: Principal Investigator, Edward ChokeTieng Chek, Senior Consultant, Vascular Service, Sengkang General Hospital
Other Study IDs: Promus PREMIER BTK
Record Dates: First submitted 2021-09-14; First posted 2021-09-23 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Peripheral Arterial Disease; Arterial Disease; Arterial Disease of Legs
Keywords: PVD; BTK; DES; PAD; Everolimus
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with CLTI and BTK lesions planned for revascularization: The study population will be CLTI patients presenting with lower limb tissue loss (ulcer or gangrene) and BTK lesions who are candidates for revascularization for limb salvage.
  Interventions: Device: Promus PREMIER BTK DES

INTERVENTIONS:
Device: Promus PREMIER BTK DES — Collect one year data of the Promus PREMIER BTK drug eluting stent in CLTI patients

SUMMARY:
The Promus Premier below-the-knee (BTK) drug-eluting stent (DES) is specifically designed to improve BTK vessel patency rates using a platinum-chromium alloy based stent that elutes the anti-restenotic drug everolimus to inhibit neo-intimal hyperplasia. Although DES stents are considered standard of care for certain BTK lesions, there is a paucity of data on the use of DES in the contemporary BTK chronic limb threatening ischemia (CLTI) population, especially in Singapore. The aim of the Promus PREMIER BTK registry is to collect one year data of the Boston Scientific Promus PREMIER BTK DES in BTK lesions in CLTI patients.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) is an atherosclerotic condition in which chronic inflammation of the arteries may result in CLTI and ultimately limb loss without treatment. This problem is likely to worsen with the increasing global prevalence of diabetes. The arterial blockage for diabetic CLTI patients occur predominantly in the BTK arteries which are challenging to treat effectively due to the high incidence of elastic recoil and high stenosis rates after plain old balloon angioplasty (POBA) of these often calcified lesions. The additional use of BTK drug-coated balloons (DCBs) have also not demonstrated any significant improvements compared to POBA. The Boston Scientific Promus Premier BTK DES is a next generation DES specifically designed to improve BTK vessel patency using a platinum-chromium alloy-based stent that elutes everolimus. It is made with the most radiopaque biocompatible alloy available with superior axial strength, exceptional conformability, maximum fracture resistance, higher radial strength and less recoil compared to cobalt alloy stent. It also has the highest labelled post-dilatation limits compared to other stents, providing clinicians with more flexibility during procedures. Subjects will be followed up at 1 month, 3 month, 6 month and 12 month post-intervention to assess primary and secondary efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

Clinical inclusion criteria

1. Subject is 21 years or older and has signed and dated the informed consent document (ICD)
2. Subject is willing and able to comply with the study procedures, and follow-up schedule
3. Subject has chronic, symptomatic related lower limb ischemia, determined by Rutherford categories 4 to 6 in the target limb, with wound(s) confined to toes/forefoot
4. Subject is a male or non-pregnant female. If female or child-bearing potential, and if sexually active must be using, or agree to use, a medically acceptable method of birth control as confirmed by the investigator

Intraoperative inclusion criteria

1. Stenotic, restenotic or occlusive target lesion(s) located in the tibioperoneal trunk, anterior tibial, posterior tibial and/or peroneal artery(ies).
2. Target lesion(s) must be at least 4cm above the ankle joint
3. A single target lesion per vessel, in up to 2 vessels, in a single limb
4. Degree of stenosis ≥ 70% by visual angiographic assessment
5. RVD is between 2.5 - 3.75mm
6. Total target lesion length (or series of lesion segments) to be treated is ≤ 140 mm (Note: Lesion segment(s) must be fully covered with up to two DES BTK stents)
7. Target vessel(s) reconstitute(s) at or above the stenting limit zone (4cm above the ankle joint)
8. Target lesion(s) is in an area that may be stented without blocking access to patent main branches
9. Treatment of all above the knee inflow lesion(s) is successful prior to treatment of the target lesion
10. Guidewire has successfully crossed the target lesion(s)

Exclusion Criteria:

Clinical exclusion criteria

1. Life expectancy ≤ 1year
2. Stroke ≤ 90 days prior to the procedure date
3. Prior or planned major amputation in the target limb
4. Previous surgery in the target vessel(s) (including prior ipsilateral crural bypass)
5. Previously implanted stent in the target vessel(s)
6. Failed PTA of target lesion/vessel ≤ 60 days prior to the procedure date
7. Heel gangrene
8. Subject has a platelet count ≤ 50 or ≥ 600 X 103/µL ≤ 30 days prior to the procedure date
9. NYHA class IV heart failure
10. Subject has symptomatic coronary artery disease (i.e., unstable angina)
11. History of myocardial infarction or thrombolysis ≤ 90 days prior to the procedure date
12. Non-atherosclerotic disease resulting in occlusion (e.g., embolism, Buerger's disease, vasculitis)
13. Subject is currently taking Canagliflozin
14. Body Mass Index (BMI) <18
15. Active septicaemia or bacteraemia
16. Coagulation disorder, including hypercoagulability
17. Contraindication to anticoagulation or antiplatelet therapy
18. Known allergies to stent or stent components
19. Known allergy to contrast media that cannot be adequately pre-medicated prior to the interventional procedure
20. Known hypersensitivity to heparin
21. Subject is on a high dose of steroids or is on immunosuppressive therapy
22. Subject is currently participating, or plans to participate in, another investigational study that may confound the results of this study

Intraoperative exclusion criteria

1. Angiographic evidence of intra-arterial acute/subacute thrombus or presence of atheroembolism
2. Treatment required in > 2 target vessels (Note: a target lesion originating in one vessel and extending into another vessel is considered 1 target vessel)
3. Treatment requires the use of alternate therapy in the target vessel(s)/lesion(s), (e.g., atherectomy, cutting balloon, re-entry devices, laser, radiation therapy)
4. Aneurysm is present in the target vessel(s)
5. Extremely calcified lesions
6. Failure to obtain <30% residual stenosis in a pre-existing lesion

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with critical limb threatening ischemia (CLTI) and below the knee (BTK) lesions planned for revascularization
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-08-16 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Number of participants with primary patency at 6 months post-procedure using duplex ultrasound | 6 months
  Primary patency using duplex ultrasound
Number of participants with major adverse events (MAE) at 6 months post-procedure | 6 months
  MAE is defined as above ankle amputation in index limb; major re-intervention; and perioperative 30-day mortality

SECONDARY OUTCOMES:
Number of participants with primary and assisted primary patency | 6 and 12 months
  Target lesion patency rate measured by duplex ultrasound
Number of participants with clinically driven target lesion revascularization | 1, 3, 6 and 12 months
  Any surgical or percutaneous intervention to the target lesion after the index procedure
Major amputation rates | 1, 3, 6 and 12 months
  Rates of amputation of the lower limb at the ankle level or above
Subject quality-of-life values by change in EQ-5D | 1, 3, 6 and 12 months
  The EQ-5D is a descriptive system of health related quality-of-life states consisting of 5 dimensions (mobility, self-care, usual activities, pain/ discomfort, anxiety/ depression) each of which can take 1 of 5 responses. The responses record 5 levels of severity (no problems / slight problems / moderate problems / severe problems / extreme problems) within a particular EQ-5D dimension. The levels are assigned a numeric code 1-5 (e.g., 1 = no problem and 5 = extreme problems). Sub score are not applicable.
Wound assessment | 1, 3, 6 and 12 months
  Descriptive characteristic of wound healing will be recorded
Change in Rutherford classification | 3, 6 and 12 months
  Change in Rutherford classification as assessed by investigator
Number of adverse events (AEs) | 1, 3, 6 and 12 months
  Adverse events (AEs) to be classified as major, serious, non-serious unanticipated, procedure-related, and device-related
30-day unplanned hospital readmission rate | 30-day
  Hospitalization related to Critical Limb-Threatening Ischemia (CLTI)
Number of participants with all-cause mortality | 6 and 12 months
  Telephone follow-up visit and/or medical chart review and/or publicly available records consultation for vital status
Change in hemodynamic outcomes | 6 and 12 months
  Change in ankle brachial index (ABI) and/or Toe pressure (TP)

CONTACTS AND LOCATIONS:
Overall Officials: Jia Sheng Tay, Principal Investigator — Sengkang General Hospital
Locations (1):
- Sengkang General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ipema J, Huizing E, Schreve MA, de Vries JPM, Unlu C. Editor's Choice - Drug Coated Balloon Angioplasty vs. Standard Percutaneous Transluminal Angioplasty in Below the Knee Peripheral Arterial Disease: A Systematic Review and Meta-Analysis. Eur J Vasc Endovasc Surg. 2020 Feb;59(2):265-275. doi: 10.1016/j.ejvs.2019.10.002. Epub 2019 Dec 27. PMID 31889657
- [Background] Bosiers M, Scheinert D, Peeters P, Torsello G, Zeller T, Deloose K, Schmidt A, Tessarek J, Vinck E, Schwartz LB. Randomized comparison of everolimus-eluting versus bare-metal stents in patients with critical limb ischemia and infrapopliteal arterial occlusive disease. J Vasc Surg. 2012 Feb;55(2):390-8. doi: 10.1016/j.jvs.2011.07.099. Epub 2011 Dec 14. PMID 22169682
- [Background] Romiti M, Albers M, Brochado-Neto FC, Durazzo AE, Pereira CA, De Luccia N. Meta-analysis of infrapopliteal angioplasty for chronic critical limb ischemia. J Vasc Surg. 2008 May;47(5):975-981. doi: 10.1016/j.jvs.2008.01.005. Epub 2008 Apr 18. PMID 18372148